CLINICAL TRIAL: NCT06762847
Title: Development And Durability Of Prosthetic Liner For Transtibial Amputee
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall22/757
Record Dates: First submitted 2024-12-13; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exp Group
  Interventions: Device: Use of Conventional Silicone Prosthetic Liner

INTERVENTIONS:
Device: Use of Conventional Silicone Prosthetic Liner — At this stage participant who will be fitted with a standard silicone liner typically used for transtibial prosthetics. Over a set duration, we will assess the liner's performance, particularly in terms of durability, comfort, skin health, and fit stability. Acting as the control group, this cohort will provide essential baseline data for comparison with the innovative prosthetic liner.

SUMMARY:
About 16% of the world's population suffers from physical disabilities, of which about 65% of the population experience lower limb amputations, and in lower limb about 50% face transtibial amputation and use transtibial prosthesis. The transtibial prosthetic users face many stump-related problems.

DETAILED DESCRIPTION:
As a physical interface, a prosthetic liner is commonly used as a transition material between residual limb and stiff socket to provide optimal comfort, fit, and functionality. By using a prosthetic liner, stump-related issues can be relieved, and long-term use of prosthetic devices achieved by an amputee. Prosthetic liners are so expensive due to being imported that patients can't afford them. My study aims to develop a low-cost prosthetic liner for transtibial amputees to ensure its availability and affordability for patients who need a prosthetic liner, by using material available at a local level like silicon to improve their ability to cushion and protect the residual limb from injuries induced by load-bearing normal and shear stresses. The study includes 1 sample size of 40 years of age males, Participents develop a prosthetic liner and then use it on these samples to determine liner durability and hope the results are in favor.

ELIGIBILITY:
Inclusion Criteria:

* Transtibial amputee with medium stump.
* Amputee which has been using the prosthetic leg for 3 years without prosthetic liners.
* Amputee with 40 years of age.

Exclusion Criteria:

* Any other amputees except transtibial.
* Amputees without using prosthetic devices.
* Amputees above 40 years of age.

Ages: 40 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Transtibial amputee with medium stump, using the prosthetic leg for 3 years without prosthetic liners. age should be 40 years
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Socket Comfort Score | 12 Months
  The socket comfort score is a numerical rating scale used to assess the comfort of a prosthetic. the score ranges from 0 to 10, with 0 being the least comfortable and 10 being the most comfortable.
Timed Up and Go (TUG) | 12 months
  This test measures the Time in seconds; lower scores indicate better performance the lower the time is the better the score is.
Skin Irritation Scale | 12 months
  Skin Irritation Scale deals with the skin irritation (Scores: 0-4, where 0 = no irritation and 4 = severe irritation)
6-Minute Walk Test | 12 months
  6-Minute Walk Test in this test we mesuares the Distance in meters; higher distance indicates better performance

CONTACTS AND LOCATIONS:
Locations (1):
- PAK Rehabilitation Centre, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No